CLINICAL TRIAL: NCT07128719
Title: Study Effects of Preoperative Modafinil on Recovery Profile of Morbidly Obese Patients Scheduled for Bariatric Surgery
Brief Title: Study Effects of Preoperative Modafinil on Recovery Profile of Morbidly Obese Patients Scheduled for Bariatric Surgery if it Can Enhance Recovery From Anesthesia
Acronym: modafinil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, foad farouk mohamed, lecturer of anesthesia, ICU and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FAMSU MS 412/2023
Record Dates: First submitted 2025-07-29; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Obese Adolescents; Bariatric Surgery
Keywords: bariatric surgery; obesity; modafinil; recovery from anethesia
MeSH Terms: conditions — Obesity | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 patients received modafinil preoperatively (Active Comparator): assessing enhancement of recovery from anesthesia
  Interventions: Drug: Modafinil
- 10 patients didnot receive modafinil preoperatively (Placebo Comparator)
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — dose of modafinil preoperatively for for active comparator

SUMMARY:
study Effects of Preoperative Modafinil on Recovery Profile of Morbidly Obese Patients Scheduled for Bariatric Surgery if it Can Enhance Recovery From Anesthesia and provide improvement in recovery

DETAILED DESCRIPTION:
The study was conducted to 20 patients scheduled for bariatric surgeries. The study group (Modafinil group) received oral 200 mg modafinil 8 hours before surgery and then another 200 mg 2 hours before surgery. The other group (Placebo group) were given placebo through the same regimen as Modafinil. Immediate recovery time, cognitive recovery, emotional (general) status, discharge from PACU according to modified Aldrete score were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 to 60 years.
2. Patients ASA II or III undergoing elective bariatric surgery.
3. BMI 30-50 kg/m2.

Exclusion Criteria:

1. Patient's refusal.
2. Age below 18 or above 60y.
3. History of cardiac disease.
4. History or known allergy to Modafinil.
5. Underlying liver or renal failure.
6. Chronic neurological or psychiatric condition.
7. Hemodynamically unstable patients.
8. History of drug dependance.
9. Habitual coffee consumption exceeding 2 cups per day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
both groups were assessed as regard incidence of enhancement of immediate and cognitive recovery Comparison between groups as regard words recall as part of cognitive recovery data. | 1 day
  Groups were compared in the primary outcome of our work (immediate recovery data) in OR by time intervals (T1, T2, T3 and T4) Comparison between groups as regard orientation as part of cognitive recovery score

SECONDARY OUTCOMES:
assessment of difference of general and emotional status between both patients groups postoperatively | 24 hours
  Groups were compared in assessment of general status and emotion and assessment of modified Aldrete score in PACU and compare between both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR